CLINICAL TRIAL: NCT02547675
Title: An Expanded Access Protocol of Oral Rociletinib (CO-1686) as Epidermal Growth Factor Receptor (EGFR)-Directed Therapy for Patients With EGFR-Mutant Non-Small Cell Lung Cancer (NSCLC) With the T790M Resistance Mutation
Brief Title: Rociletinib (CO-1686) USA Expanded Access Program
Status: No longer available | Type: Expanded Access
Sponsor: Clovis Oncology, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CO-1686-031
Record Dates: First submitted 2015-09-10; First posted 2015-09-11 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — rociletinib

INTERVENTIONS:
Drug: Rociletinib — Rociletinib will be administered to patients orally
  Other Names: CO-1686

SUMMARY:
To provide access to rociletinib for patients with advanced or metastatic EGFR-mutant NSCLC who have been treated previously with EGFR directed therapy and have evidence of a T790M mutation (T790M+).

DETAILED DESCRIPTION:
This is an open-label, multi-center study in the US, which allows for expanded access to rociletinib for patients with advanced or metastatic, EGFR-mutant T790M+ NSCLC who were previously treated with at least one prior EGFR TKI therapy (≥2nd line). Patients will receive oral rociletinib twice daily on study as long as they have clinical benefit and until they have access to FDA-approved rociletinib.

ELIGIBILITY:
Key Inclusion Criteria:

* Unresectable locally advanced or metastatic NSCLC with EGFR activating mutation (excluding exon 20 insertion) and presence of the T790M mutation
* Prior treatment with an approved or experimental EGFR-directed therapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Adequate hematological and biological function
* Written informed consent on an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved ICF before any study-specific evaluation

Key Exclusion Criteria:

* Eligibility for other enrolling clinical trials of rociletinib
* Leptomeningeal carcinomatosis or other untreated or symptomatic CNS metastases (asymptomatic CNS metastases allowed if clinically stable without requirement for steroid dose increase for at least 4 weeks)
* History of prior interstitial lung disease
* Concurrent use of QT-prolonging medication
* Cardiac abnormalities:

  * Clinically significant abnormal 12-lead ECG, QT interval corrected using Fridericia's method (QTcF) > 450 ms
  * Inability to measure QT interval on ECG
  * Personal or family history of long QT syndrome
  * Implantable pacemaker or implantable cardioverter defibrillator
  * Resting bradycardia < 55 beats/min
* Presence of serious or unstable concomitant systemic disorder incompatible with the clinical study (eg, substance abuse, uncontrolled intercurrent illness including active infection, arterial thrombosis, symptomatic pulmonary embolism, and other active malignancy associated with life expectancy of less than 1 year)
* Pregnant or breastfeeding females and male or female patients who refuse to use adequate contraception during the study and for 12 weeks after the last dose of rociletinib
* Any contraindication, allergy, or hypersensitivity to rociletinib or excipients

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Compassionate Care Research Group, Inc., Fountain Valley, California
  - Pacific Cancer Care, Monterey, California
  - Sutter Cancer Institute, Sacramento, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Halifax Health - Center for Oncology, Daytona Beach, Florida
  - UF Health Center Orlando, Orlando, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Billings Clinic, Billings, Montana
  - Tulsa Cancer Institute, Tulsa, Oklahoma